CLINICAL TRIAL: NCT02692820
Title: Preventing Preterm Birth With Probiotics - Pilot Randomised Trial
Brief Title: Preventing Preterm Birth With Probiotics
Acronym: PrePro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 010294QM
Record Dates: First submitted 2015-09-28; First posted 2016-02-26 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-01

CONDITIONS: Preterm Birth
Keywords: Preterm; Probiotic
MeSH Terms: conditions — Premature Birth | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Experimental): Those who provide consent will be randomised to receive once daily for the remainder of their pregnancy capsules of probiotics (containing Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 (each at 2.5 x 109 colony forming units (CFUs)). The product contains freeze-dried bacteria and excipients in a gelatin capsule.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Those who provide consent will be randomised to receive once daily for the remainder of their pregnancy capsules of the placebo containing excipients alone in a gelatin capsule
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Probiotic — The probiotic capsule contains the two probiotics Lactobacillus rhamnosus GR-1 (GR-1) and Lactobacillus reuteri RC-14 (RC-14). The product contains freeze-dried bacteria and excipients in a gelatin capsule;
  Arms: Probiotic
Other: Placebo Comparator — The placebo contains excipients alone in a gelatin capsule
  Arms: Placebo

SUMMARY:
Babies born preterm (before completing 37 weeks in the womb) are at increased risk of long-term disability and death. The investigators do not fully understand the cause(s) of preterm birth but it occurs more frequently when the normal, healthy bacteria (called Lactobacilli) in a woman's birth canal are replaced with unhealthy bacteria. Previous attempts to get rid of the unhealthy bacteria with antibiotics have not shown to affect the risk of preterm birth. The reason for this may be that what is required is the replacement of Lactobacilli in the birth canal. This can be done by asking women to take capsules containing lactobacilli once daily. To study whether oral Lactobacilli capsules compared with dummy capsules can reduce the risk of preterm birth, a large study involving approximately 10,000 women would be required. But the investigators do not know whether women would agree to take part in and complete such a study, and this is what the investigators wish to study in the small, initial study described here. The results of this study will show whether probiotics produce the desired biological effects on vaginal bacteria, and whether it would be feasible to perform the larger, definitive study of their effectiveness in prevention of preterm birth.

DETAILED DESCRIPTION:
Preterm birth (PTB) is defined as the birth of a baby before the completion of 37 weeks gestation in the womb. It is the major cause of infant mortality particularly during the first month of life. Approximately 75 per cent of babies who die during the first 28 days of life are born before 37 weeks gestation. Survivors of PTB are at increased risk of long-term disabilities such as cerebral palsy, sight and hearing impairment, learning and behavioural problems, epilepsy, and hospital readmissions. Even late preterm births, defined as PTB at 34--36 weeks gestation, which account for 70% of all preterm births in England and Wales, are at increased risk of death and disability compared with babies born at term. Although the prevalence of adverse long--term outcome is highest among children born at the earliest gestational ages, the much higher number of births at 34--36 weeks of gestation compared with earlier gestations means that this group of children makes a major contribution to the number of children adversely affected. PTB and its consequences can have negative emotional and psychosocial impacts on parents and families.

In addition to its impact on individuals and families, the financial consequences for the public sector of caring for children born preterm are significant. The cost of care up to the age of 18 for children born preterm has been estimated to exceed £3 billion per year in England and Wales at 2006 prices. It has been estimated that a hypothetical intervention that delayed PTB by 1 week across all gestational age categories would reduce the public sector cost of PTB by £1 billion annually.

About one third of PTBs occur because early delivery is indicated due to complications in the mother or the unborn baby (fetus); the remaining two thirds occur spontaneously. The rate of PTB has increased by 19% from 1990 to 2010 in developed countries. At the same time, there has been a marked improvement in the survival rates of PTBs but a similar reduction in adverse outcomes has not been seen. Thus, the absolute numbers of individuals adversely affected is increasing.

Infection within the womb (intrauterine infection) is strongly associated with spontaneous PTB. The commonest pathway for intrauterine infection is the ascent of unhealthy bacteria from the vagina and cervix into the womb. Bacterial vaginosis (BV), in which the normally dominant healthy bacteria in the vagina (lactobacilli) are replaced with unhealthy bacteria, is strongly associated with PTB. Lactobacilli, principally the strains that produce higher levels of the chemical hydrogen peroxide, appear to protect against BV and reduce the risk of PTB.

Despite substantial evidence linking BV with PTB, the results of trials of antibiotic treatment of BV in pregnancy have not produced clear evidence of benefit. The reason for this might be that it is not the eradication of unhealthy bacteria that is required but rather the replacement of unhealthy bacteria with the normally dominant lactobacilli. One way of achieving this could be by administering lactobacilli-containing capsules (probiotics) to pregnant women. Oral probiotics taken during pregnancy may directly alter the vaginal bacteria and in so doing protect the cervical opening from ascending infection.

The investigators have formally reviewed the medical literature on the use of probiotics to prevent PTB. There is some evidence from medical trials which suggests that probiotics taken during pregnancy can reduce the risk of PTB but the trials have either been too small or of poor quality for the results to be conclusive. The results of an observational study on nearly 19,000 pregnant women suggested that probiotic- containing foods reduced the risk of spontaneous PTB.

The best way to determine whether probiotics can reduce the risk of PTB is by performing a type of study called a double-blind, randomised controlled trial (RCT). In such a trial, the participants are allocated to receive either probiotic supplements or dummy (placebo) supplements. The allocation to a particular supplement is purely by chance (random) and neither the participants nor the researchers know the allocation of any participant until the end of the trial (double-blind). Then, by looking at the difference in the rate of PTB between the groups it would be possible to say whether probiotics can reduce the rate of PTB. The investigators have estimated that an RCT that could detect a useful difference in the rate of PTB between the two groups would require the participation of approximately 10,000 women and cost several million pounds. Given that approximately 20,000 deliveries occur annually in inner North East London alone, there are sufficient women in this region who would be eligible for participation in such a RCT. However, the willingness of women to participate in and complete such a trial is unknown.

A small, pilot trial is required to determine what proportion of pregnant women would participate in a probiotics and PTB trial and the proportion that would complete the study. The proposal here, the PrePro trial, is designed to gather these data which will inform the feasibility, planning and execution of a large RCT looking at the effects of probiotics on PTB.

Potential risks and benefits of probiotics The World Health Organisation defines probiotics as live micro-organisms that confer a health benefit on the host when administered in adequate amounts. They can displace and kill pathogens, and modulate the immune response by interfering with the inflammatory cascade that can cause preterm labour. Administration of probiotics by mouth or intravaginally is safe and effective in reducing the incidence of or treating urogenital infections. There is no evidence of adverse consequences for mothers or their infants as a result of probiotic exposure during pregnancy. Acceptability of and compliance with daily ingestion of probiotic or placebo for a few weeks during mid-pregnancy was found to be high. The particular probiotic strains proposed for this study have been shown to be acceptable to and safe in pregnant women, and can colonise the vagina within 4 weeks of commencing oral intake.

A large intervention trial of ingesting oral capsules from early pregnancy to the end of gestation has not been performed in the UK. For such a trial to be successful, it is essential to gather data that will inform its feasibility, planning and execution. PrePro is designed to provide these data. This trial will be conducted in compliance with the study protocol, relevant regulations, and the MRC Guidelines for Good Clinical Practice (GCP).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 16 years and over at the time of the booking appointment.
* Women who are between 9-14 weeks gestation at the time of the dating scan.

Exclusion Criteria:

* Lack of informed, written consent

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2016-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The microbiological effect of the probiotic on the vaginal flora during pregnancy, | 18 months
  To evaluate the microbiological effects of probiotics on vaginal flora the investigators will compare treatments groups regarding the proportion of women with bacterial vaginosis (BV) at delivery and the proportion of women with vaginal colonisation with intervention strains at delivery.
The proportion of eligible women recruited into the trial | 18 months
  The primary analysis will also involve the estimation of the proportions of the primary outcomes (i.e. eligible women recruited into the trial, recruited women who complete the trial and adhere to the intervention treatment until delivery).
The proportions of recruited women who complete the trial and adhere to the intervention until delivery | 18 months
  The primary analysis will also involve the estimation of the proportions of the primary outcomes (i.e. eligible women recruited into the trial, recruited women who complete the trial and adhere to the intervention treatment until delivery).

SECONDARY OUTCOMES:
Questionnaire/interview assessment of reasons for participation and non-participation, trial attrition, and non-adherence to trial protocol by ethnic groups (subject to funding) | 18 months
  Subject to receipt of additional funding, a qualitative sub-study will examine the acceptability to women of using probiotics as a dietary supplement during pregnancy and participation in the trial, and the fidelity to treatment allocation. Methods will include direct observation of recruitment episodes and recorded interviews with participants and non-participants by a qualitative social researcher. Qualitative data analysis will use a framework approach supported by the use of dedicated software
Core outcomes for use in studies on preterm birth prevention from case report forms | 18 months
  This is defined as new-born outcome before or at first discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Khalid S Khan, Phd, Principal Investigator — Queen Mary University of London; Rehan Khan, MD, Principal Investigator — Barts Health NHS
Locations (2):
- United Kingdom (2):
  - Barts Health NHS Trust, London
  - Homerton University Hospital, London

REFERENCES:
- [Background] Office for National Statistics, (2014a). Gestation-specific Infant Mortality in England and Wales, 2012 tables. [Internet] Available at: http://www.ons.gov.uk/ons/rel/child-health/gestation-specific-infant-mortality-in-england-and-wales/2012/rft-table-1.xls
- [Background] Doyle LW, Ford G, Davis N. Health and hospitalistions after discharge in extremely low birth weight infants. Semin Neonatol. 2003 Apr;8(2):137-45. doi: 10.1016/S1084-2756(02)00221-X. PMID 15001150
- [Background] Arpino C, Compagnone E, Montanaro ML, Cacciatore D, De Luca A, Cerulli A, Di Girolamo S, Curatolo P. Preterm birth and neurodevelopmental outcome: a review. Childs Nerv Syst. 2010 Sep;26(9):1139-49. doi: 10.1007/s00381-010-1125-y. Epub 2010 Mar 27. PMID 20349187
- [Background] Boyle JD, Boyle EM. Born just a few weeks early: does it matter? Arch Dis Child Fetal Neonatal Ed. 2013 Jan;98(1):F85-8. doi: 10.1136/archdischild-2011-300535. Epub 2011 Aug 24. PMID 21865487
- [Background] Saigal S, Doyle LW. An overview of mortality and sequelae of preterm birth from infancy to adulthood. Lancet. 2008 Jan 19;371(9608):261-9. doi: 10.1016/S0140-6736(08)60136-1. PMID 18207020
- [Background] Mangham LJ, Petrou S, Doyle LW, Draper ES, Marlow N. The cost of preterm birth throughout childhood in England and Wales. Pediatrics. 2009 Feb;123(2):e312-27. doi: 10.1542/peds.2008-1827. PMID 19171583
- [Background] Goldenberg RL, Hauth JC, Andrews WW. Intrauterine infection and preterm delivery. N Engl J Med. 2000 May 18;342(20):1500-7. doi: 10.1056/NEJM200005183422007. No abstract available. PMID 10816189
- [Background] Blencowe H, Cousens S, Oestergaard MZ, Chou D, Moller AB, Narwal R, Adler A, Vera Garcia C, Rohde S, Say L, Lawn JE. National, regional, and worldwide estimates of preterm birth rates in the year 2010 with time trends since 1990 for selected countries: a systematic analysis and implications. Lancet. 2012 Jun 9;379(9832):2162-72. doi: 10.1016/S0140-6736(12)60820-4. PMID 22682464
- [Background] Office for National Statistics, (2014b). Childhood, Infant and Perinatal Mortality in England and Wales, 2012. [Internet] Available at: http://www.ons.gov.uk/ons/rel/vsob1/child-mortality-statistics--childhood--infant-and-perinatal/2012/rft-cms-2012.xls
- [Background] Costeloe KL, Hennessy EM, Haider S, Stacey F, Marlow N, Draper ES. Short term outcomes after extreme preterm birth in England: comparison of two birth cohorts in 1995 and 2006 (the EPICure studies). BMJ. 2012 Dec 4;345:e7976. doi: 10.1136/bmj.e7976. PMID 23212881
- [Background] Guaschino S, De Seta F, Piccoli M, Maso G, Alberico S. Aetiology of preterm labour: bacterial vaginosis. BJOG. 2006 Dec;113 Suppl 3:46-51. doi: 10.1111/j.1471-0528.2006.01122.x. PMID 17206964
- [Background] Donders GG, Van Calsteren K, Bellen G, Reybrouck R, Van den Bosch T, Riphagen I, Van Lierde S. Predictive value for preterm birth of abnormal vaginal flora, bacterial vaginosis and aerobic vaginitis during the first trimester of pregnancy. BJOG. 2009 Sep;116(10):1315-24. doi: 10.1111/j.1471-0528.2009.02237.x. Epub 2009 Jun 17. PMID 19538417
- [Background] Hawes SE, Hillier SL, Benedetti J, Stevens CE, Koutsky LA, Wolner-Hanssen P, Holmes KK. Hydrogen peroxide-producing lactobacilli and acquisition of vaginal infections. J Infect Dis. 1996 Nov;174(5):1058-63. doi: 10.1093/infdis/174.5.1058. PMID 8896509
- [Background] Wilks M, Wiggins R, Whiley A, Hennessy E, Warwick S, Porter H, Corfield A, Millar M. Identification and H(2)O(2) production of vaginal lactobacilli from pregnant women at high risk of preterm birth and relation with outcome. J Clin Microbiol. 2004 Feb;42(2):713-7. doi: 10.1128/JCM.42.2.713-717.2004. PMID 14766841
- [Background] Mosbah A, Mesbah MR. (2009) A study of the role of hydrogen peroxide production by lactobacilli in preterm labor. Int J Med Med Sci, 1:388-95.
- [Background] Brocklehurst P, Gordon A, Heatley E, Milan SJ. Antibiotics for treating bacterial vaginosis in pregnancy. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD000262. doi: 10.1002/14651858.CD000262.pub4. PMID 23440777
- [Background] Cooper NA, Moores R; East London Preterm Prevention Collaboration. A review of the literature regarding nutritional supplements and their effect on vaginal flora and preterm birth. Curr Opin Obstet Gynecol. 2014 Dec;26(6):487-92. doi: 10.1097/GCO.0000000000000126. PMID 25379767
- [Background] Othman M, Neilson JP, Alfirevic Z. Probiotics for preventing preterm labour. Cochrane Database Syst Rev. 2007 Jan 24;2007(1):CD005941. doi: 10.1002/14651858.CD005941.pub2. PMID 17253567
- [Background] Unlu C, Donders G. Use of lactobacilli and estriol combination in the treatment of disturbed vaginal ecosystem: a review. J Turk Ger Gynecol Assoc. 2011 Dec 1;12(4):239-46. doi: 10.5152/jtgga.2011.57. eCollection 2011. PMID 24592002
- [Background] Zhao T-F, Zhong L, Luo D.(2010) Living preparation of lactobacillus versus metronidazole for bacterial vaginosis in pregnancy: a systematic review. Chin J Evid-based Med, 10:1338-44.
- [Background] Myhre R, Brantsaeter AL, Myking S, Gjessing HK, Sengpiel V, Meltzer HM, Haugen M, Jacobsson B. Intake of probiotic food and risk of spontaneous preterm delivery. Am J Clin Nutr. 2011 Jan;93(1):151-7. doi: 10.3945/ajcn.110.004085. Epub 2010 Oct 27. PMID 20980489
- [Background] Yeganegi M, Watson CS, Martins A, Kim SO, Reid G, Challis JR, Bocking AD. Effect of Lactobacillus rhamnosus GR-1 supernatant and fetal sex on lipopolysaccharide-induced cytokine and prostaglandin-regulating enzymes in human placental trophoblast cells: implications for treatment of bacterial vaginosis and prevention of preterm labor. Am J Obstet Gynecol. 2009 May;200(5):532.e1-8. doi: 10.1016/j.ajog.2008.12.032. Epub 2009 Mar 14. PMID 19285652
- [Background] Dugoua JJ, Machado M, Zhu X, Chen X, Koren G, Einarson TR. Probiotic safety in pregnancy: a systematic review and meta-analysis of randomized controlled trials of Lactobacillus, Bifidobacterium, and Saccharomyces spp. J Obstet Gynaecol Can. 2009 Jun;31(6):542-552. doi: 10.1016/S1701-2163(16)34218-9. PMID 19646321
- [Background] Lindsay KL, Brennan L, McAuliffe FM. Acceptability of and compliance with a probiotic capsule intervention in pregnancy. Int J Gynaecol Obstet. 2014 Jun;125(3):279-80. doi: 10.1016/j.ijgo.2014.01.004. Epub 2014 Feb 19. No abstract available. PMID 24636629
- [Background] Krauss-Silva L, Moreira ME, Alves MB, Braga A, Camacho KG, Batista MR, Almada-Horta A, Rebello MR, Guerra F. A randomised controlled trial of probiotics for the prevention of spontaneous preterm delivery associated with bacterial vaginosis: preliminary results. Trials. 2011 Nov 8;12:239. doi: 10.1186/1745-6215-12-239. PMID 22059409
- [Background] Reid G, Charbonneau D, Erb J, Kochanowski B, Beuerman D, Poehner R, Bruce AW. Oral use of Lactobacillus rhamnosus GR-1 and L. fermentum RC-14 significantly alters vaginal flora: randomized, placebo-controlled trial in 64 healthy women. FEMS Immunol Med Microbiol. 2003 Mar 20;35(2):131-4. doi: 10.1016/S0928-8244(02)00465-0. PMID 12628548
- [Derived] Davidson SJ, Barrett HL, Price SA, Callaway LK, Dekker Nitert M. Probiotics for preventing gestational diabetes. Cochrane Database Syst Rev. 2021 Apr 19;4(4):CD009951. doi: 10.1002/14651858.CD009951.pub3. PMID 33870484
- [Derived] Husain S, Allotey J, Drymoussi Z, Wilks M, Fernandez-Felix BM, Whiley A, Dodds J, Thangaratinam S, McCourt C, Prosdocimi EM, Wade WG, de Tejada BM, Zamora J, Khan K, Millar M. Effects of oral probiotic supplements on vaginal microbiota during pregnancy: a randomised, double-blind, placebo-controlled trial with microbiome analysis. BJOG. 2020 Jan;127(2):275-284. doi: 10.1111/1471-0528.15675. Epub 2019 Apr 1. PMID 30932317